CLINICAL TRIAL: NCT03526627
Title: Advanced Care Management in Patients With Advanced Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201711101RIND
Record Dates: First submitted 2018-03-06; First posted 2018-05-16 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-05

CONDITIONS: Advanced Heart Failure
Keywords: advanced care management, advanced heart failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient with advanced heart failure: we included the patients with advanced heart failure who had the poor cardiac function(LVEF<=30%) and was admitted to the general ward or emergency room within one year.

SUMMARY:
The purpose of this study is to explore the trajectory of advanced management care in patients with heart failure over a period of 9 months, then comparing the medical treatment accepted by patients after 2 years later and compliance with the preferences of patients and their families.

DETAILED DESCRIPTION:
this study is to observe the trajectory of the advanced care management on patients with advanced heart failure and follow the difference between the actual medical treatment accepted by patients on 2years later and the preference of the patient and their families.

the advance care management in this study is mean the patients who know about the preference of medical treatment, communication, and prognosis of illness. we also measure the sense of coherence, self-efficacy and their quality of life to compare their relationship of the advanced care management.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with AHA stage D, or NYHA class function 4, or LVEF<=30%.
* has one or more than one symptoms such as dyspnea, lower legs edema, weakness.
* ever admission to the hospital (include emergency room or the general room)

Exclusion Criteria:

* with other end-stage diseases such cancer, dementia, COPD, ESRD...etc.
* had other physical, cognitive, or psychological condition which may influence their answer.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patient with advanced heart disease and received medical treatment now.
Sampling Method: Non-Probability Sample
Enrollment: 227 (Estimated)
Dates: Start 2018-01-04 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
advanced care management | 3 months for each interval and 4 times on each patient (total 9 months on this study)
  we use a modified questionnaire "assessment the medical needs and preference on terminal patients and their families (Tang, et al., 2004) by literature review and named "The prognosis and message status on patients with advanced Heart failure. the questionnaire include 3 parts: medical preference in their advanced status, communication between physician and patients and physician and their families ( the definition of families in this study is the major medical decision for the patients), and the knowledge of disease prognosis. The questionnaire include 17 items with continue and category variables. Before study we use expert validity from 5 experts who works in group at least 10 years. Each items is scored on a five-point Likert scale range from 0(not at all) to 4 (very appropriate to this study). The overall score was calculated as the average of all items and finally we got 3.67-points.

CONTACTS AND LOCATIONS:
Overall Officials: Kai-di Kao, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng, Taiwan